CLINICAL TRIAL: NCT03647956
Title: Atezolizumab in Combination With Bevacizumab, Carboplatin and Pemetrexed for EGFR-mutant Metastatic Non-small Cell Lung Cancer Patients After Failure of EGFR Tyrosine Kinase Inhibitors: a Single Arm Phase 2 Study
Brief Title: Atezolizumab in Combination With Bevacizumab, Carboplatin and Pemetrexed for EGFR-mutant Metastatic NSCLC Patients After Failure of EGFR Tyrosine Kinase Inhibitors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML40560
Record Dates: First submitted 2018-08-24; First posted 2018-08-27 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: NSCLC Stage IIIB; NSCLC Stage IV; EGFR Activating Mutation
Keywords: Atezolizumab; Bevacizumab; Carboplatin; Pemetrexed; EGFR-mutant metastatic NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Bevacizumab; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Using Atezolizumab, a PD-L1 inhibitor, in combination with bevacizumab, carboplatin and pemetrexed to treat patients with EGFR mutated, advanced non-small cell lung cancer (NSCLC) after failure of EGFR tyrosine kinase inhibitors.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab (trade name Tecentriq) is a fully humanized, engineered monoclonal antibody of IgG1 isotype against the protein programmed cell death-ligand 1 (PD-L1).
  Other Names: Tecentriq
Drug: Bevacizumab — Bevacizumab is a recombinant humanized monoclonal antibody that blocks angiogenesis by inhibiting vascular endothelial growth factor A (VEGF-A).
  Other Names: Avastin
Drug: Carboplatin — Carboplatin, sold under the trade name Paraplatin among others, is a chemotherapy medication used to treat a number of forms of cancer.
  Other Names: Paraplatin
Drug: Pemetrexed — Pemetrexed (brand name Alimta) is a chemotherapy drug manufactured and marketed by Eli Lilly and Company. Its indications are the treatment of pleural mesothelioma and non-small cell lung cancer.
  Other Names: Alimta

SUMMARY:
This project will recruit 40 EGFR-mutant metastatic non-small cell lung cancer patients who failed any EGFR tyrosine kinase inhibitors.

All recruited patients will receive 1200mg Azetolizumab administered over 60 minutes (1st cycle) and 30 minutes (2nd cycle onwards) intravenously, as well as 7.5mg/kg bevacizumab administered over 90 minutes (1st cycle), 60 minutes (2nd cycle) and 30 minutes (3rd cycle onwards) for every 3 weeks, until radiographically documented disease progression, unacceptable toxicity as judged by investigators or patient withdrawal.

The primary objective is to assess the progression-free survival of this treatment population, and to identify potential genomic and immunologic biomarkers for treatment response. Objective response rate (ORR) will be the primary efficacy endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Stage IIIB or IV NSCLC with known EGFR activating mutation not amenable to curative surgery or radiotherapy.
* Radiological documentation of disease progression following one or more lines of EGFR TKI treatment but have not received palliative chemotherapy. For tumors with uncommon EGFR mutation, including exon 20 insertions, exon 18 point mutations and or complex mutations, patients should have received one or more lines of EGFR TKI treatment.
* Patients must receive tumor EGFR genotyping by peripheral blood circulating tumor-DNA (ctDNA)
* Measurable disease as defined by RECIST 1.1 Criteria.
* At least 18 years of age.
* World Health Organisation (WHO) performance status 0-2 with no deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks
* At least one lesion, not previously irradiated and not chosen for biopsy during the study screening period, that can be accurately measured at baseline as ≥ 10mm in the longest diameter (except lymph nodes which must have short axis ≥ 15mm) with computerised tomography (CT) or magnetic resonance imaging (MRI) which is suitable for accurate repeated measurements.
* Normal bone marrow and organ function as defined below:
* Marrow: Hemoglobin ≥10.0 gm/dL, absolute granulocyte count (AGC) ≥1,000/mm3 platelets ≥100,000/mm3, absolute lymphocyte count ≥1000/mm3.
* Hepatic: Serum/plasma total bilirubin ≤1.5 x upper limit of normal (ULN) with the exception of <2.9 mg/dL for patients with Gilbert's disease, ALT (SGPT) and AST (SGOT) ≤2.5 x ULN.
* Renal: Serum/plasma creatinine (sCr) ≤1.5 x upper limit of normal, or creatinine clearance (Ccr) ≥50 mL/min.
* Serum/plasma albumin > 3.0 gm/dL
* For female patients of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception that results in a low failure rate (< 1% per year) when used consistently and correctly, and to continue its use for 5 months after the last dose of atezolizumab and/or 6 months after the last dose of bevacizumab. Such methods include: combined (estrogen and progestogen containing) hormonal contraception, progestogen-only hormonal contraception associated with inhibition of ovulation together with another additional barrier method always containing a spermicide, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner (on the understanding that this is the only one partner during the whole study duration), and sexual abstinence.
* Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Previous exposure to platinum-based palliative chemotherapy. The use of neoadjuvant or adjuvant platinum-based chemotherapy more than 6 months before study enrollment is allowed
* Previous exposure to VEGF inhibitor for anti-cancer treatment
* Prior treatment with any other anti-programmed cell death protein-1 (anti-PD-1), or PD Ligand-1 (PD-L1) or PD Ligand-2 (PDL2) agent or an antibody targeting other immuno-regulatory receptors or mechanisms
* Patients carries EGFR genotype T790M but have not received 3rd generation EGFR TKI Osimertinib
* Currently participating or has participated in a study of an investigational agent or using an investigational device within 4 weeks of administration of atezolizumab
* Expected to require any other form of antineoplastic therapy while on study
* Patients with untreated symptomatic brain metastases. Patients with treated brain metastases will be allowed if brain imaging obtained greater than 7 days from trial enrollment reveals stable disease. Patients with small (< 3mm) asymptomatic brain metastasis are allowed to enroll. Patients on steroids doses higher than 10 mg of prednisone (or its equivalent) are excluded
* Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for > 2 weeks prior to randomization
* Leptomeningeal disease
* Uncontrolled tumor-related pain
* Patients requiring pain medication must be on a stable regimen at study entry.
* Symptomatic lesions amenable to palliative radiotherapy (e.g., bone metastases or metastases causing nerve impingement) should be treated prior to randomization. Patients should be recovered from the effects of radiation. There is no required minimum recovery period.
* Asymptomatic metastatic lesions whose further growth would likely cause functional deficits or intractable pain (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for locoregional therapy, if appropriate, prior to randomization.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Patients with indwelling catheters (e.g., PleurX®) are allowed. Uncontrolled or symptomatic hypercalcemia (> 1.5 mmol/L ionized calcium or Ca > 12 mg/dL or corrected serum calcium > ULN). Patients who are receiving denosumab prior to randomization must be willing and eligible to receive a bisphosphonate instead while in the study.
* Malignancies other than NSCLC within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death (e.g., expected 5-year OS > 90%) treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous-cell skin cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent)
* On chronic systemic steroid therapy or on any other form of immunosuppressive medication
* Has received a live-virus vaccination within 30 days of planned treatment start
* Clinically active diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction, or abdominal carcinomatosis (known risks factors for bowel perforation)
* Severe hypersensitivity reaction to treatment with another monoclonal antibody (mAb)
* Active autoimmune disease that has required systemic treatment in the past 2 years (replacement therapies for hormone deficiencies are allowed)
* Systemic cytotoxic chemotherapy, antineoplastic biologic therapy, or major surgery within 3 weeks of the first dose of study medication
* Active infection requiring therapy
* History of Human Immunodeficiency Virus (HIV)
* Hepatitis B carrier: Patients with HBV infection were required to be receiving effective antiviral therapy and have a viral load less than 100 IU/mL at screening
* Active Hepatitis C
* Interstitial lung disease or pneumonitis requiring oral or IV glucocorticoids
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study
* Psychiatric disorders and substance (drug/alcohol) abuse

Exclusion Criteria Related to Bevacizumab

* Inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg). Anti-hypertensive therapy to achieve these parameters is allowable.
* Prior history of hypertensive crisis or hypertensive encephalopathy
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to randomization
* History of hemoptysis (≥ one-half teaspoon of bright red blood per episode) within 1 month prior to randomization
* Evidence of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation)
* Current or recent (within 10 days of randomization) use of aspirin (> 325 mg/day) or treatment with dipyramidole, ticlopidine, clopidogrel, and cilostazol
* Current use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes that has not been stable for > 2 weeks prior to randomization
* The use of full-dose oral or parenteral anticoagulants is permitted as long as the INR or aPTT is within therapeutic limits (according to the medical standard of the enrolling institution) and the patient has been on a stable dose of anticoagulants for at least 2 weeks prior to randomization.
* Prophylactic anticoagulation for the patency of venous access devices is allowed, provided the activity of the agent results in an INR < 1.5 × ULN and aPTT is within normal limits within 14 days prior to randomization.
* Prophylactic use of low-molecular-weight heparin (i.e., enoxaparin 40 mg/day) is permitted.
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to the first dose of bevacizumab
* History of abdominal or tracheosphageal fistula or gastrointestinal perforation within 6 months prior to randomization
* Clinical signs of gastrointestinal obstruction or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding
* Evidence of abdominal free air not explained by paracentesis or recent surgical procedure
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Proteinuria, as demonstrated by urine dipstick or > 1.0 g of protein in a 24-hour urine collection
* All patients with ≥ 2 + protein on dipstick urinalysis at baseline must undergo a 24-hour urine collection and must demonstrate ≤

  1 g of protein in 24 hours.
* Known sensitivity to any component of bevacizumab
* Clear tumor infiltration into the thoracic great vessels is seen on imaging
* Clear cavitation of pulmonary lesions is seen on imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-04-03 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 3 years
  The percentage of patients with radiologically complete or partial response as determined by the investigator according to RECIST version 1.1.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | 3 years
  PFS is measured from the date of study enrollment to radiographically documented progression according to RECIST 1.1 or death from any cause (whichever occurs first).
  Participants alive and without disease progression or lost to follow-up will be censored at the date of their last radiographic assessment.
Time to progression (TTP) | 3 years
  TTP is measured from the date of study enrollment to radiographically documented progression according to RECIST 1.1. This does not include death from any cause.
Duration of response (DoR) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tai-Chung Lam, FRCR, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Clinical Oncology, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lynch TJ, Bell DW, Sordella R, Gurubhagavatula S, Okimoto RA, Brannigan BW, Harris PL, Haserlat SM, Supko JG, Haluska FG, Louis DN, Christiani DC, Settleman J, Haber DA. Activating mutations in the epidermal growth factor receptor underlying responsiveness of non-small-cell lung cancer to gefitinib. N Engl J Med. 2004 May 20;350(21):2129-39. doi: 10.1056/NEJMoa040938. Epub 2004 Apr 29. PMID 15118073
- [Background] Shi Y, Au JS, Thongprasert S, Srinivasan S, Tsai CM, Khoa MT, Heeroma K, Itoh Y, Cornelio G, Yang PC. A prospective, molecular epidemiology study of EGFR mutations in Asian patients with advanced non-small-cell lung cancer of adenocarcinoma histology (PIONEER). J Thorac Oncol. 2014 Feb;9(2):154-62. doi: 10.1097/JTO.0000000000000033. PMID 24419411
- [Background] Mok TS, Wu YL, Thongprasert S, Yang CH, Chu DT, Saijo N, Sunpaweravong P, Han B, Margono B, Ichinose Y, Nishiwaki Y, Ohe Y, Yang JJ, Chewaskulyong B, Jiang H, Duffield EL, Watkins CL, Armour AA, Fukuoka M. Gefitinib or carboplatin-paclitaxel in pulmonary adenocarcinoma. N Engl J Med. 2009 Sep 3;361(10):947-57. doi: 10.1056/NEJMoa0810699. Epub 2009 Aug 19. PMID 19692680
- [Background] Maemondo M, Inoue A, Kobayashi K, Sugawara S, Oizumi S, Isobe H, Gemma A, Harada M, Yoshizawa H, Kinoshita I, Fujita Y, Okinaga S, Hirano H, Yoshimori K, Harada T, Ogura T, Ando M, Miyazawa H, Tanaka T, Saijo Y, Hagiwara K, Morita S, Nukiwa T; North-East Japan Study Group. Gefitinib or chemotherapy for non-small-cell lung cancer with mutated EGFR. N Engl J Med. 2010 Jun 24;362(25):2380-8. doi: 10.1056/NEJMoa0909530. PMID 20573926
- [Background] Zhou C, Wu YL, Chen G, Feng J, Liu XQ, Wang C, Zhang S, Wang J, Zhou S, Ren S, Lu S, Zhang L, Hu C, Hu C, Luo Y, Chen L, Ye M, Huang J, Zhi X, Zhang Y, Xiu Q, Ma J, Zhang L, You C. Erlotinib versus chemotherapy as first-line treatment for patients with advanced EGFR mutation-positive non-small-cell lung cancer (OPTIMAL, CTONG-0802): a multicentre, open-label, randomised, phase 3 study. Lancet Oncol. 2011 Aug;12(8):735-42. doi: 10.1016/S1470-2045(11)70184-X. Epub 2011 Jul 23. PMID 21783417
- [Background] Sequist LV, Yang JC, Yamamoto N, O'Byrne K, Hirsh V, Mok T, Geater SL, Orlov S, Tsai CM, Boyer M, Su WC, Bennouna J, Kato T, Gorbunova V, Lee KH, Shah R, Massey D, Zazulina V, Shahidi M, Schuler M. Phase III study of afatinib or cisplatin plus pemetrexed in patients with metastatic lung adenocarcinoma with EGFR mutations. J Clin Oncol. 2013 Sep 20;31(27):3327-34. doi: 10.1200/JCO.2012.44.2806. Epub 2013 Jul 1. PMID 23816960
- [Background] Yu HA, Arcila ME, Rekhtman N, Sima CS, Zakowski MF, Pao W, Kris MG, Miller VA, Ladanyi M, Riely GJ. Analysis of tumor specimens at the time of acquired resistance to EGFR-TKI therapy in 155 patients with EGFR-mutant lung cancers. Clin Cancer Res. 2013 Apr 15;19(8):2240-7. doi: 10.1158/1078-0432.CCR-12-2246. Epub 2013 Mar 7. PMID 23470965
- [Background] Janne PA, Yang JC, Kim DW, Planchard D, Ohe Y, Ramalingam SS, Ahn MJ, Kim SW, Su WC, Horn L, Haggstrom D, Felip E, Kim JH, Frewer P, Cantarini M, Brown KH, Dickinson PA, Ghiorghiu S, Ranson M. AZD9291 in EGFR inhibitor-resistant non-small-cell lung cancer. N Engl J Med. 2015 Apr 30;372(18):1689-99. doi: 10.1056/NEJMoa1411817. PMID 25923549
- [Background] Yang CJ, Tsai MJ, Hung JY, Liu TC, Chou SH, Lee JY, Hsu JS, Tsai YM, Huang MS, Chong IW. Pemetrexed had significantly better clinical efficacy in patients with stage IV lung adenocarcinoma with susceptible EGFR mutations receiving platinum-based chemotherapy after developing resistance to the first-line gefitinib treatment. Onco Targets Ther. 2016 Mar 16;9:1579-87. doi: 10.2147/OTT.S100164. eCollection 2016. PMID 27051298
- [Background] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Background] Brahmer JR, Tykodi SS, Chow LQ, Hwu WJ, Topalian SL, Hwu P, Drake CG, Camacho LH, Kauh J, Odunsi K, Pitot HC, Hamid O, Bhatia S, Martins R, Eaton K, Chen S, Salay TM, Alaparthy S, Grosso JF, Korman AJ, Parker SM, Agrawal S, Goldberg SM, Pardoll DM, Gupta A, Wigginton JM. Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012 Jun 28;366(26):2455-65. doi: 10.1056/NEJMoa1200694. Epub 2012 Jun 2. PMID 22658128
- [Background] Akbay EA, Koyama S, Carretero J, Altabef A, Tchaicha JH, Christensen CL, Mikse OR, Cherniack AD, Beauchamp EM, Pugh TJ, Wilkerson MD, Fecci PE, Butaney M, Reibel JB, Soucheray M, Cohoon TJ, Janne PA, Meyerson M, Hayes DN, Shapiro GI, Shimamura T, Sholl LM, Rodig SJ, Freeman GJ, Hammerman PS, Dranoff G, Wong KK. Activation of the PD-1 pathway contributes to immune escape in EGFR-driven lung tumors. Cancer Discov. 2013 Dec;3(12):1355-63. doi: 10.1158/2159-8290.CD-13-0310. Epub 2013 Sep 27. PMID 24078774
- [Background] Chen N, Fang W, Zhan J, Hong S, Tang Y, Kang S, Zhang Y, He X, Zhou T, Qin T, Huang Y, Yi X, Zhang L. Upregulation of PD-L1 by EGFR Activation Mediates the Immune Escape in EGFR-Driven NSCLC: Implication for Optional Immune Targeted Therapy for NSCLC Patients with EGFR Mutation. J Thorac Oncol. 2015 Jun;10(6):910-23. doi: 10.1097/JTO.0000000000000500. PMID 25658629
- [Background] Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, Ready NE, Chow LQ, Vokes EE, Felip E, Holgado E, Barlesi F, Kohlhaufl M, Arrieta O, Burgio MA, Fayette J, Lena H, Poddubskaya E, Gerber DE, Gettinger SN, Rudin CM, Rizvi N, Crino L, Blumenschein GR Jr, Antonia SJ, Dorange C, Harbison CT, Graf Finckenstein F, Brahmer JR. Nivolumab versus Docetaxel in Advanced Nonsquamous Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Oct 22;373(17):1627-39. doi: 10.1056/NEJMoa1507643. Epub 2015 Sep 27. PMID 26412456
- [Background] Herbst RS, Baas P, Kim DW, Felip E, Perez-Gracia JL, Han JY, Molina J, Kim JH, Arvis CD, Ahn MJ, Majem M, Fidler MJ, de Castro G Jr, Garrido M, Lubiniecki GM, Shentu Y, Im E, Dolled-Filhart M, Garon EB. Pembrolizumab versus docetaxel for previously treated, PD-L1-positive, advanced non-small-cell lung cancer (KEYNOTE-010): a randomised controlled trial. Lancet. 2016 Apr 9;387(10027):1540-1550. doi: 10.1016/S0140-6736(15)01281-7. Epub 2015 Dec 19. PMID 26712084
- [Background] Rittmeyer A, Barlesi F, Waterkamp D, Park K, Ciardiello F, von Pawel J, Gadgeel SM, Hida T, Kowalski DM, Dols MC, Cortinovis DL, Leach J, Polikoff J, Barrios C, Kabbinavar F, Frontera OA, De Marinis F, Turna H, Lee JS, Ballinger M, Kowanetz M, He P, Chen DS, Sandler A, Gandara DR; OAK Study Group. Atezolizumab versus docetaxel in patients with previously treated non-small-cell lung cancer (OAK): a phase 3, open-label, multicentre randomised controlled trial. Lancet. 2017 Jan 21;389(10066):255-265. doi: 10.1016/S0140-6736(16)32517-X. Epub 2016 Dec 13. PMID 27979383
- [Background] Gainor JF, Shaw AT, Sequist LV, Fu X, Azzoli CG, Piotrowska Z, Huynh TG, Zhao L, Fulton L, Schultz KR, Howe E, Farago AF, Sullivan RJ, Stone JR, Digumarthy S, Moran T, Hata AN, Yagi Y, Yeap BY, Engelman JA, Mino-Kenudson M. EGFR Mutations and ALK Rearrangements Are Associated with Low Response Rates to PD-1 Pathway Blockade in Non-Small Cell Lung Cancer: A Retrospective Analysis. Clin Cancer Res. 2016 Sep 15;22(18):4585-93. doi: 10.1158/1078-0432.CCR-15-3101. Epub 2016 May 25. PMID 27225694
- [Background] Jiang L, Su X, Zhang T, Yin X, Zhang M, Fu H, Han H, Sun Y, Dong L, Qian J, Xu Y, Fu X, Gavine PR, Zhou Y, Tian K, Huang J, Shen D, Jiang H, Yao Y, Han B, Gu Y. PD-L1 expression and its relationship with oncogenic drivers in non-small cell lung cancer (NSCLC). Oncotarget. 2017 Apr 18;8(16):26845-26857. doi: 10.18632/oncotarget.15839. PMID 28460468
- [Background] Ahn MJ, Sun JM, Lee SH, Ahn JS, Park K. EGFR TKI combination with immunotherapy in non-small cell lung cancer. Expert Opin Drug Saf. 2017 Apr;16(4):465-469. doi: 10.1080/14740338.2017.1300656. Epub 2017 Mar 8. PMID 28271729
- [Background] Hata A, Katakami N, Nanjo S, Okuda C, Kaji R, Masago K, Fujita S, Yoshida H, Zama K, Imai Y, Hirata Y. Programmed death-ligand 1 expression according to epidermal growth factor receptor mutation status in pretreated non-small cell lung cancer. Oncotarget. 2017 Dec 1;8(69):113807-113816. doi: 10.18632/oncotarget.22837. eCollection 2017 Dec 26. PMID 29371947
- [Background] Tseng YH, Hung HY, Sung YC, Tseng YC, Lee YC, Whang-Peng J, Chen YM. Efficacy of chemotherapy in epidermal growth factor receptor (EGFR) mutated metastatic pulmonary adenocarcinoma patients who had acquired resistance to first-line EGFR tyrosine kinase inhibitor (TKI). J Chemother. 2016;28(1):50-8. doi: 10.1179/1973947815Y.0000000027. PMID 25976428
- See also: Overview of Hong Kong Cancer Statistics of 2014. — http://www3.ha.org.hk/cancereg/pdf/overview/Summary%20of%20CanStat%202014.pdf